CLINICAL TRIAL: NCT05954130
Title: The Effect of Web-Based Education Specific to Sexual Health During Pregnancy on Sexual Life
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Sule Gokyildiz Surucu, Prof., Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 04.11.2022/38
Record Dates: First submitted 2023-06-06; First posted 2023-07-20 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Sexual Behavior
Keywords: pregnancy, sexual life, education
MeSH Terms: conditions — Sexual Behavior | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: experimental and control
Who Masked: Participant
Masking Description: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Application Support Specific to Sexual Health in Pregnancy (Experimental): The training module will consist of 3 sessions. The first session will last 1 hour, with 45 minutes of interactive lecture and 15 minutes of question and answer. The second and third sessions will last 1 hour, with 45 minutes of interactive narration and 15 minutes of qualitative interviews. Module sessions will have a dynamic structure that takes into account the needs of the pregnant woman in her trimester. The content of the training sessions will be structured on the following topics.
  Interventions: Other: Education
- control (No Intervention): No training will be given to the pregnant women in the control group who accepted to participate in the study.

INTERVENTIONS:
Other: Education — Sexual Health in Pregnancy
  Arms: Mobile Application Support Specific to Sexual Health in Pregnancy

SUMMARY:
Pregnancy is an important process with many changes in a woman's life. During this period, the sexual lives of couples may be affected due to anatomical, physiological and psychological changes. While sexual intercourse during pregnancy strengthens the harmony between spouses, emotional bond, and self-confidence of the woman, its role is important in terms of the continuation of the marriage.

The development of technology in the world and in our country has led to an increase in the use of mobile devices. The emergence of telehealth and mobile applications with the Covid-19 pandemic has enabled individuals to access information whenever they want and more easily.

The aim of this study was to determine the effect of mobile application support given to pregnant women for sexual health on sexual function and quality of sexual life.

It is planned to develop a mobile application in this direction by preparing a guide, with the foresight that sexuality during pregnancy is not an easily expressed subject and that pregnant women and health workers need training materials. After the power analysis, it is aimed to reach a total of 70 people, 35 in the experimental group and 35 in the control group. Data will be collected with Personal Information Form, Female Sexual Function Index, Sexual Life Quality Scale and Qualitative Interview Form.

Based on the developed guide and mobile application, training will be given to pregnant women in the first, second and third trimesters, and it is thought that the mobile application support specific to sexual health during pregnancy may contribute to increasing sexual function and sexual life quality.

DETAILED DESCRIPTION:
This thesis study was designed to determine the effect of mobile application support given to pregnant women for sexual health on sexual function and quality of sexual life. In this thesis, it is planned to develop a mobile application in this direction by preparing a guide, with the foresight that sexuality during pregnancy is not an easily expressed subject and that pregnant women and health workers need training materials on this subject. Based on the developed guide and mobile application, it is thought that by providing continuous training to pregnant women, it can contribute to increasing women's sexual function and sexual life quality.

Research Hypotheses

* H0 a: Mobile application support for sexual health during pregnancy has no effect on sexual function.
* H1 a: Mobile application support specific to sexual health during pregnancy has an effect on sexual function.
* H0 b: The mobile application support for sexual health during pregnancy has no effect on the quality of sexual life.
* H1 b: Mobile application support specific to sexual health during pregnancy has an effect on the quality of sexual life.

ELIGIBILITY:
Inclusion Criteria:

* In the first 3 months of pregnancy
* Speaks and understands Turkish
* Being able to read and write
* Not having received prior education about sexuality during pregnancy

Exclusion Criteria:

* Having a risky pregnancy (under 18 years of age, having a chronic and psychiatric disease, etc.)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — will be applied to pregnant women
Enrollment: 70 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index | Change in sexual functions during pregnancy at 9 months
  It was developed as a 19-item multidimensional scale to evaluate female sexual function. The scale assesses sexual problems or function in the last 4 weeks. In the structure of the scale; There are 6 sub-dimensions: desire, arousal, lubrication (lubrication, wetting), orgasm, satisfaction and pain. Each item is scored from zero to 5. Accordingly, the highest raw score that can be obtained from the scale is 95.0, and the lowest raw score is 4.0.

SECONDARY OUTCOMES:
Sexual Quality of Life Scale | Change in the quality of sexual life in 9 months of pregnancy
  The scale is easy to apply, six-point Likert type, which individuals can answer on their own, and consists of 18 items. It is expected that each item will be answered considering his sexual life in the last four weeks. In scoring the scale, each question is scored between 1-6. In this system, it will be scored as (1=Strongly Agree, 2=Strongly Agree, 3=Partly Agree, 4=Somewhat Disagree, 5=Strongly Agree, 6=Strongly Disagree). In this way, the range of points that can be obtained from the scale is between 18-108.

CONTACTS AND LOCATIONS:
Overall Officials: Şule GÖKYILDIZ SÜRÜCÜ, Prof., Study Director — gokyildizsule@gmail.com; Emel SALCAN, Msc.Midwife, Principal Investigator — emelers@hotmail.com
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)